CLINICAL TRIAL: NCT01836237
Title: The Use of Wound Protectors to Prevent Surgical Site Infection for Whipples (Pancreatoduodenectomy) With Intrabiliary Stents: A Randomized Controlled Trial.
Brief Title: The Use of Wound Protector in Whipple's Procedure With Intrabiliary Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Chad G. Ball, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E - 24807
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Surgical Wound Infection; Pancreatic Neoplasms
Keywords: Surgical site infection rate; Wound protector use; Whipple
MeSH Terms: conditions — Surgical Wound Infection; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alexis group (Experimental): In experimental group patients, the surgeon will use Alexis - a wound protector during surgery.
  Interventions: Device: Alexis - a wound protector
- Control group (No Intervention): In no intervention group patients, the surgeon will not use any wound protector during surgery.

INTERVENTIONS:
Device: Alexis - a wound protector — Alexis is a double ring, self-retaining circumferential device that is designed to protect incision site during surgical manipulation.
  Arms: Alexis group

SUMMARY:
Background: There are no published studies regarding the use of wound protectors in the context of surgical site infection (SSI) rates among patients receiving a pancreatoduodenectomy (Whipple) with preoperatively placed intrabiliary stents. In high volume experiences, the SSI rate is 40-50% within this cohort. In Calgary, preoperative biliary stent placement for bile duct decompression represents the norm given typical surgical wait times. In addition to having higher associated lengths of hospital stay, ICU admissions, hospital re-admissions, and overall mortality, patients with SSI are also delayed, and often omitted, in their progression to critical oncologic adjuvant chemotherapy. As a result, SSI remain crucial and devastating complications for pancreas surgeons and their patients alike.

Methods: The investigators will complete a randomized controlled trial evaluating the rate of SSI in adult patients who undergo a pancreatoduodenectomy following biliary stent placement when wound protectors are employed versus no wound protector use. This trial will employ block randomization. All four University of Calgary Heapato-Pancreatico-Biliary (HPB) surgeons will participate with a planned inclusion of all patients scheduled to undergo a pancreatoduodenectomy.

Analysis: The investigators will use an intention to treat approach to the analysis. Categorical baseline data will be analyzed using the Fisher exact probability test. Non-categorical baseline data will be analyzed using the Student t test. SSI rates will be determined using the Fisher exact probability test.

Hypothesis: Wound protectors will reduce the SSI rate in patients undergoing a pancreatoduodenectomy with preoperatively placed intrabiliary stents.

Potential Impact: Given the tremendous oncologic, economic, and psychological impact of SSI following pancreatoduodenectomy, the epidemic incidence of this complication must be reduced. The additional crippling effect of refusing (Medicare) payment for any patient who receives a SSI in the United States has launched all techniques and analyses that can potentially reduce this complication into the National health care agenda. In Canada, health care utilization and economics are always a relevant and ever expanding area of importance. It is crucial that the investigators reduce complications such as SSI, regardless of individual payer sources.

DETAILED DESCRIPTION:
Introduction

The Department of Surgery at the University of Calgary has a long and proud tradition of research surrounding surgical site infections (SSI). More specifically, former surgeon and Department Chair Dr. Peter Cruse prospectively studied 23,649 surgical wounds following operative intervention. This massive study remains unmatched in size by a single institution publication. Dr. Cruse and Ms. Rosemary Foord demonstrated a decrease in SSI rates with the pre-surgical use of hexachlorophene wash and by not shaving the surgical site1. They observed an increase in SSI rates with advanced age, use of drains, prolonged hospital stay before the operation, and longer operative times. Dr. Cruse is directly responsible for confirming the validity of the wound classification system currently in use throughout the world (clean, clean-contaminated, contaminated, and dirty). We propose to carry on the tradition of this line of investigation, reinforcing Calgary as a world leader in SSI research.

SSI are a frequent and costly source of post-operative morbidity. They are the most common complication following gastrointestinal and biliary tract surgery, occurring in 5-30% of patients. SSI are associated with a two-fold increased risk of in-hospital mortality, a 50% increase in intensive care admission, a 6-day mean increase in hospital stay, and a five-fold increased rate of readmission. SSI also have additional and highly negative consequences in the treatment of oncology patients. More specifically, medical oncologists wait until all operative wounds are entirely healed prior to beginning adjuvant chemotherapy. This delay is both oncologically concerning, as well as psychologically destructive to highly stressed patients with poor associated survivals. Furthermore, with a significant SSI, this delay often leads to a total omission of adjuvant therapies as a whole. The estimated increased cost per SSI ranges from $1,300 to $5,000 in the United States. In Canada, a 1998 study estimated $3,937 per infection, resulting from increased hospital stay, as well as emergency department and clinic visits. The implications of these costs have now become paramount given that both U.S. Medicare and Medicaid currently deny any reimbursement for patients who obtain an SSI while admitted to hospital. In addition, patients who develop SSI experience psychosocial distress, loss of income, and loss of productivity. Prevention of SSI is therefore a vitally important goal in delivering quality care to patients. The SSI rate is 40-50% in patients undergoing pancreatoduodenectomy with intrabiliary stents, the population of interest for this study.

Wound protectors are devices designed to protect the abdominal wound tissue edges from contamination and trauma during laparotomy. A major reason for their conception and use is a theoretical reduction in risk of SSI. Various devices with similar intent have been described since the 1960s, falling into two main design categories: (1) Those with an internal and external ring connected by impervious plastic, and (2) Those with a single, internal ring connected to a drape which extends outward, over the wound edges and onto the abdomen where they are affixed with adhesive or clips.A recent meta-analysis of randomized controlled trials was conducted by a team led by the Principal Investigator to evaluate whether impervious plastic wound protectors reduce the risk of surgical site infection following gastrointestinal and biliary surgery. Six studies representing 1,008 patients were included. Wound protectors were associated with a 45% decrease in SSI (p = 0.04). The Alexis Wound Protector, a ring based model, had evidence of superiority to other products and has been selected for this study based on this finding.

Methods

Recruitment: Contact information for study candidates will be obtained by the project's research fellow from the offices of the participating (4) surgeons. Patients will be contacted prior to their surgery by the research fellow and will be provided information regarding the study. Patients who consent to participate will be randomized.

Randomization process: This study is a simple, two-arm randomized clinical trial (RCT) with block randomization. Allocation will be concealed before the patient enters study. Patients will be randomized by the Research fellow following consent. Allocation will be provided to surgeon in a sealed envelope to be opened immediately before surgery. Patients and the data analyst will be blind to allocation; the surgeons cannot be blinded. Charts will be blinded for data abstraction.

Data collection: Information will be collected by chart review from the operative report and patient records by the research fellow in the Department of Surgery.

Data elements to be collected include:

Date of birth, Sex, American Society of Anesthesiologist (ASA) score, Surgeon, Site (if more than one facility), Fellow/resident/clerk present (y/n), Surgical procedure, Antibiotic prophylaxis received (y/n) and time given, Information about repeat antibiotic prophylaxis (for longer surgeries), Antibiotic type/combination, Type of wound protector and manufacturer, Prep type (ETOH based, chlorhexidine based, iodine based), Hair removal, Medications given, Packing, Drains, Wound classification, Wound closure technique & dressing type, Length of surgery, Surgical suite infection control factors (e.g. UV, OR ventilation) if these differ, Transfusions,

Patient records:

Current use of corticosteroids/immune suppressant, Preoperative chemotherapy, Smoking history, Co-morbidities (diabetes, hypertension, etc.), Body Mass Index (BMI).

The presence of an SSI will be determined according to guidelines developed by the Centers for Disease Control. More specifically, SSI is defined as being the presence of at least one of the following:

1. Purulent drainage, with or without laboratory conformation, from the superficial incision.
2. Organisms isolated from an aseptically obtained culture of fluid from the superficial incision.
3. At least one of the following signs or symptoms of infection:

   pain or tenderness, localized swelling, redness and superficial incision is deliberately opened by surgeon, unless incision is culture-negative.
4. Diagnosis of superficial incisional SSI by the surgeon or attending physician.

Analysis

We will use an intention to treat approach to the analysis to avoid the effects of crossover and dropout. To achieve a power (superiority trial) of 90%, and alpha of 0.05 with a 5% crossover and a 40% expected SSI rate in control versus 10% in wound protector groups, the total sample size is 78 (i.e. 39 in each arm).

Resources

This project will capitalize on an existing research team who can work collaboratively with the Principal Investigator and research assistant to carry out the project effectively and efficiently. The current research team includes a clinical research fellow with experience recruiting research participants from this patient population and a project manager who can assist with ethics applications, manuscript writing and reporting. Additionally, the Principal Investigator will benefit from mentorship by an experienced investigator who can provide guidance not only on methodology, interpretation of data and publication strategies, but also on the day-to-day logistics of running a research project.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years or older, undergoing pancreatoduodenectomy with intrabiliary stents in place at Foothills Medical centre, Calgary, Alberta.

Exclusion Criteria:

* Patients will be excluded if they have had long-term steroid use or are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) Rate | 1 month
  SSI will be evaluated on a daily basis by residents, the research/clinical fellow and/or Hepato-Pancreatico-Biliary Team by visual inspection of each wound.

CONTACTS AND LOCATIONS:
Overall Officials: Chad G. Ball, MD, Principal Investigator — University of Calgary, Calgary, Alberta, Canada
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] Cruse PJ, Foord R. A five-year prospective study of 23,649 surgical wounds. Arch Surg. 1973 Aug;107(2):206-10. doi: 10.1001/archsurg.1973.01350200078018. No abstract available. PMID 4719566
- [Background] Murray BW, Huerta S, Dineen S, Anthony T. Surgical site infection in colorectal surgery: a review of the nonpharmacologic tools of prevention. J Am Coll Surg. 2010 Dec;211(6):812-22. doi: 10.1016/j.jamcollsurg.2010.07.025. Epub 2010 Oct 25. No abstract available. PMID 20980173
- [Background] Horiuchi T, Tanishima H, Tamagawa K, Matsuura I, Nakai H, Shouno Y, Tsubakihara H, Inoue M, Tabuse K. Randomized, controlled investigation of the anti-infective properties of the Alexis retractor/protector of incision sites. J Trauma. 2007 Jan;62(1):212-5. doi: 10.1097/01.ta.0000196704.78785.ae. PMID 17215757
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Dimick JB, Chen SL, Taheri PA, Henderson WG, Khuri SF, Campbell DA Jr. Hospital costs associated with surgical complications: a report from the private-sector National Surgical Quality Improvement Program. J Am Coll Surg. 2004 Oct;199(4):531-7. doi: 10.1016/j.jamcollsurg.2004.05.276. PMID 15454134
- [Background] Zhan C, Miller MR. Excess length of stay, charges, and mortality attributable to medical injuries during hospitalization. JAMA. 2003 Oct 8;290(14):1868-74. doi: 10.1001/jama.290.14.1868. PMID 14532315
- [Background] Zoutman D, McDonald S, Vethanayagan D. Total and attributable costs of surgical-wound infections at a Canadian tertiary-care center. Infect Control Hosp Epidemiol. 1998 Apr;19(4):254-9. doi: 10.1086/647804. PMID 9605274
- [Background] Reid K, Pockney P, Draganic B, Smith SR. Barrier wound protection decreases surgical site infection in open elective colorectal surgery: a randomized clinical trial. Dis Colon Rectum. 2010 Oct;53(10):1374-80. doi: 10.1007/DCR.0b013e3181ed3f7e. PMID 20847618
- [Background] Paquette IM, Swenson BR, Kwaan MR, Mellgren AF, Madoff RD. Thirty-day outcomes in patients treated with en bloc colectomy and pancreatectomy for locally advanced carcinoma of the colon. J Gastrointest Surg. 2012 Mar;16(3):581-6. doi: 10.1007/s11605-011-1691-7. Epub 2011 Sep 29. PMID 21956432
- [Background] Kimura F, Shimizu H, Yoshidome H, Ohtsuka M, Kato A, Yoshitomi H, Nozawa S, Furukawa K, Mitsuhashi N, Sawada S, Takeuchi D, Ambiru S, Miyazaki M. Increased plasma levels of IL-6 and IL-8 are associated with surgical site infection after pancreaticoduodenectomy. Pancreas. 2006 Mar;32(2):178-85. doi: 10.1097/01.mpa.0000202959.63977.5c. PMID 16552338
- [Background] Lee P, Waxman K, Taylor B et al. Use of wound-protection system and postoperative wound-infection rates in open appendectomy. Arch Surg 2009; 144:872-875.
- [Background] Edwards JP, Ho AL, Tee MC, Dixon E, Ball CG. Wound protectors reduce surgical site infection: a meta-analysis of randomized controlled trials. Ann Surg. 2012 Jul;256(1):53-9. doi: 10.1097/SLA.0b013e3182570372. PMID 22584694
- [Background] Sookhai S, Redmond HP, Deasy JM. Impervious wound-edge protector to reduce postoperative wound infection: a randomised, controlled trial. Lancet. 1999 May 8;353(9164):1585. doi: 10.1016/S0140-6736(99)00950-2. No abstract available. PMID 10334259
- [Background] Gamble SS, Hopton DS. Plastic ring wound drapes in elective colorectal surgery. J R Coll Surg Edinb. 1984 Jul;29(4):232-3. No abstract available. PMID 6384492
- [Background] Katthagen BD, Zamani P, Jung W. [Effect of surgical draping on bacterial contamination in the surgical field]. Z Orthop Ihre Grenzgeb. 1992 May-Jun;130(3):230-5. doi: 10.1055/s-2008-1040144. German. PMID 1642040
- [Derived] Bressan AK, Roberts DJ, Edwards JP, Bhatti SU, Dixon E, Sutherland FR, Bathe O, Ball CG. Efficacy of a dual-ring wound protector for prevention of incisional surgical site infection after Whipple's procedure (pancreaticoduodenectomy) with preoperatively-placed intrabiliary stents: protocol for a randomised controlled trial. BMJ Open. 2014 Aug 21;4(8):e005577. doi: 10.1136/bmjopen-2014-005577. PMID 25146716